CLINICAL TRIAL: NCT07249268
Title: Comparative Diagnostic Yield of Contrast-Enhanced Versus Conventional Ultrasound Guidance for Coaxial Biopsy of Hepatic Lesions: A Propensity Score-Matched Analysis
Brief Title: Comparative Diagnostic Yield of Contrast-Enhanced Versus Conventional Ultrasound Guidance for Coaxial Biopsy of Hepatic Lesions
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Lijuan Yan, Principal Investigator, The First Affiliated Hospital of Xiamen University
Other Study IDs: XMFHIIT-2025SL218
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Hepatic Lesions
Keywords: Liver Biopsy; Focal Liver Lesion; Coarse Needle Biopsy; Contrast-enhanced Ultrasound; Coaxial Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CEUS Group: CEUS-guided coaxial biopsy for hepatic lesions
  Interventions: Procedure: CEUS or Contrast enhanced Ultrasound
- US Group: US-guided coaxial biopsy for hepatic lesions
  Interventions: Procedure: US

INTERVENTIONS:
Procedure: CEUS or Contrast enhanced Ultrasound — CEUS-guided coaxial biopsy for hepatic lesions
  Groups: CEUS Group
Procedure: US — US-guided coaxial biopsy for hepatic lesions
  Groups: US Group

SUMMARY:
This study compared two methods used to guide needle biopsies of suspicious lumps (lesions) in the liver. A biopsy is a procedure where a small sample of tissue is taken to make a diagnosis. Doctors often use standard ultrasound (US) to see the lesion and guide the needle. Another method uses a special dye (contrast agent) injected into a vein during the ultrasound, which is called contrast-enhanced ultrasound (CEUS). The dye helps blood vessels and the lesion "light up" on the screen. The researchers wanted to find out if using CEUS leads to a more successful biopsy than using standard US alone.

DETAILED DESCRIPTION:
This study compared two different methods used to guide needles during a percutaneous (through the skin) biopsy of a focal liver lesion (a suspicious mass or lump in the liver). The goal was to see if one method was better than the other at ensuring a successful and diagnostic biopsy.

The researchers looked back at the records of 330 patients who had a liver biopsy. Of these, 113 had a CEUS-guided biopsy and 217 had a standard US-guided biopsy. To ensure a fair comparison, they used a statistical method to create two perfectly matched groups of 92 patients each. The patients in these groups were very similar in terms of factors like the size and location of their liver lesion, so that the only major difference was the type of guidance used (CEUS or US).

For most patients with a liver lesion that can be seen on a standard ultrasound, this study suggests that using the more advanced and expensive CEUS method does not increase the chances of a successful biopsy. The standard ultrasound guidance is just as effective.

Therefore, the routine use of CEUS for all liver biopsies may not be necessary. This helps in managing healthcare resources wisely. However, CEUS remains a valuable tool for specific situations where a lesion is very difficult to see clearly on a standard ultrasound scan. Doctors can reserve CEUS for these more challenging cases.

ELIGIBILITY:
Inclusion Criteria:

* Indeterminate liver lesions on prior imaging (CT/MRI).
* Coaxial biopsy performed with 18G introducer needle.

Exclusion Criteria:

* Coagulopathy (INR >1.5, platelets <50×109/L).
* Contraindications to ultrasound contrast agents.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients underwent CEUS-guided or conventional US-guided coaxial biopsy for focal hepatic lesions.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
the biopsy success rate | from enrollment to the end of the biopsy
  the biopsy success rate of liver lesion

SECONDARY OUTCOMES:
vasovagal reaction | during the procedure
  A vasovagal reaction is a sudden drop in your heart rate and blood pressure. This reduces blood flow to your brain, which can cause you to feel dizzy, sweaty, and nauseous, and can sometimes lead to fainting.
bleeding | during the procedure
  bleeding due to biopsy
pneumothorax | during the procedure
  A pneumothorax (often called a collapsed lung) happens when air leaks into the space between your lung and your chest wall.
shock | during the procedure
  Shock is a critical state of circulatory failure where the body's organs are starved of oxygen due to low blood flow, which can be caused by severe bleeding, heart failure, major infection, or a severe allergic reaction.
unplanned hospitalization | 48 hours after the surgery
  An unplanned hospitalization is an urgent admission to a hospital, typically through the emergency department, for an unexpected and serious medical event or a sudden worsening of a pre-existing condition.
death | 48 hours after the surgery
  Death is the permanent and irreversible end of all life functions in a living organism.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ultrasound, The First Affiliated Hospital of Xiamen University, 55 Zhenhai Road, Xiamen, China, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No